CLINICAL TRIAL: NCT06290817
Title: A Prospective, Multicenter, Single-arm Clinical Study on the Treatment of Newly Diagnosed Diffuse Large B-cell Lymphoma With High-risk of CNS Relapse Defined by CNS-IPI Using Orelabrutinib in Combination With R-CDOP Regimen
Brief Title: Orelabrutinib Combined With R-CDOP for DLBCL Patients With High-risk of CNS Relapse Defined by CNS-IPI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Huizhou Municipal Central Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Affiliated Hospital of Jiaxing University (Other); The Second Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0724
Record Dates: First submitted 2024-02-27; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib combined with R-CDOP regimen (Experimental): Participants will receive 150 mg of oral orelabrutinib once daily with R-CDOP on day 1 of each cycle (21 days)
  Interventions: Drug: Orelabrutinib combined with R-CDOP regimen

INTERVENTIONS:
Drug: Orelabrutinib combined with R-CDOP regimen — All participants were treated with the orelabrutinib combined with R-CHOP regimen (O-RCDOP). The treatment plan involved orelabrutinib tablets at 150mg QD (once daily) from day 1 to day 21, Rituximab at 375mg/m2 on day 1; Cyclophosphamide at 750mg/m2 on day 1; Liposomal Doxorubicin at 30mg/m2 on day 0; Vincristine at 25mg/m2 on day 1 (maximum dose 40mg); and Prednisone at 100mg from day 1 to day 5. The treatment cycles were set every 21 days for a total of 6-8 cycles. Dose adjustments were made for elderly patients for Cyclophosphamide and Liposomal Doxorubicin based on age: 70-80% of the dose for those aged 70-80 years old, and 50-60% of the dose for those older than 80 years.

SUMMARY:
This is a prospective, multicenter, single-arm clinical study on the treatment of newly diagnosed diffuse large B-cell lymphoma with high-risk of CNS relapse defined by CNS-IPI using Orelabrutinib in combination with R-CDOP regimen.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is an aggressive form of B-cell lymphoma, where the dual expression of Myc and BCL-2 genes in non-germinal center B-cell like (non-GCB) lymphomas is associated with a poor prognosis when treated with the standard R-CHOP regimen. Bruton's tyrosine kinase (BTK), a key kinase in the B-cell receptor (BCR) signaling pathway, is an important target for the treatment of B-cell lymphomas. Studies have shown that the first-generation BTK inhibitor Ibrutinib when combined with the R-CHOP regimen for previously untreated patients with dual-expressing, non-GCB lymphomas, can improve event-free survival rates. Orelabrutinib, as a new generation BTK inhibitor independently developed in China, possesses higher inhibitory activity against BTK kinase and can penetrate the blood-brain barrier, offering potential benefits for patients at high risk of central nervous system relapse. The novel anthracycline drug-Liposomal Doxorubicin, which has almost no cardiac toxicity, suggests that the combination of Orelabrutinib with the R-CDOP regimen could improve the adverse prognosis of DLBCL patients at high risk of central relapse. This is a prospective, multicenter, single-arm clinical study on the treatment of newly diagnosed diffuse large B-cell lymphoma with high-risk CNS-IPI using Orelabrutinib in combination with R-CDOP regimen. All participants were treated with the Orelabrutinib combined with R-CDOP regimen. The treatment cycles were set every 21 days for a total of 6-8 cycles. During the study treatment period, researchers conducted a tumor assessment (with a 1-week time window allowed) after the screening period and once again after the 4th, 6th, or 8th cycle of treatment to evaluate the antitumor efficacy of the investigational drug. After all treatment cycles were completed, follow-up visits were conducted every 3 months until the end of the 3-year period. The median duration of follow-up was 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old; ECOG score 0-3;
2. Histologically confirmed diffuse large B-cell lymphoma, including DLBCL and transformed DLBCL;
3. CNS-IPI≥4 points
4. Previously untreated participants with CD20-positive DLBCL,;
5. Heart, liver, and kidney function: creatinine < 2 times the normal upper limit (ULN); ALT (alanine aminotransferase)/AST (Aspartate Aminotransferase) < 2.5ULN; Total bilirubin < 2ULN; Cardiac ejection fraction (EF) ≥50%.
6. At least one measurable lesion.
7. Have the sufficient understanding ability and voluntarily sign informed consent.

Exclusion Criteria:

1. Patients with evidence of CNS involvement ;
2. Clinically significant active cardiovascular disease, such as uncontrolled arrhythmia, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease as determined by the New York Heart Association (NYHA) functional scale, or a history of myocardial infarction within 6 months before screening;
3. Human immunodeficiency virus (HIV) infection;
4. Pregnant or lactating women;
5. Other tumors that require treatment;
6. Uncontrolled active infection;
7. The HBV DNA copy number of active hepatitis after antiviral treatment can not be controlled within 2×103/ml.
8. unable to understand and follow the research protocol or unable to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
2-year central nervous system relapse rate | up to 2 years
  The proportion of patients with central nervous system recurrence within two years from enrollment accounted for all patients treated with drugs.

SECONDARY OUTCOMES:
Complete Response Rate | At the end of Cycle 3 and Cycle 6（each cycle is 21 days）
  The rate of patients who achieved complete response after treatment.
Overall Response Rate (ORR) | At the end of Cycle 3 and Cycle 6（each cycle is 21 days）
  The rate of patients who achieved CR or PR after treatment.
2-year Overall survival (OS) rate | Up to 2 years
  2-year overall survival (OS) rate Accessed by the investigator
1-year Overall survival (OS) rate | Up to 1 year
  1-year overall survival (OS) rate Accessed by the investigator
2-year progression-free survival (PFS) rate | 2 years after enrollment of final patient
  Number of non-progression cases/all enrolled cases at 2 years
1-year progression-free survival (PFS) rate | 1 year after enrollment of final patient
  Number of non-progression cases/all enrolled cases at 1 year
Occurrence of hematologic adverse events and non-hematologic adverse events according to CTCAE V4.03 | Up to 3 years
  The safety of Orelabrutinib is measured by the occurrence of hematologic adverse events and non-hematologic adverse events according to CTCAE V4.03

OTHER OUTCOMES:
Occurrence of adverse events and serious adverse events according to CTCAE V4.03 | Up to 3 years
  The safety of Orelabrutinib measured by the occurrence of adverse events and serious adverse events according to CTCAE V4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, Study Director — 15.1 Second affiliated hospital， School of Medicine， Zhejiang University
Locations (6):
- China (6):
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Zhejiang, Zhejiang
  - Huzhou Central Hospital, Huzhou
  - Affiliated hospital of Jiaxing University , the First Hospital of Jiaxing, Jiaxing
  - Affiliated hospital of Jiaxing University , the Second Hospital of Jiaxing, Jiaxing
  - Ningbo Medical Center LiHuili Hospital, Ningbo
  - Taizhou Hospital of Zhejiang, Taizhou